CLINICAL TRIAL: NCT03994679
Title: Feasibility and Performance of Brainlab Iplan Software, in Comparison to Freeware for Virtual Bone Graft Planning in Unilateral Cleft Patients: a Retrospective, Pilot Study
Brief Title: Feasibility and Performance of Virtual Software for Virtual Bone Graft Planning in Cleft Patients
Acronym: VIR-CLEFT
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Krisztian Nagy, principal investigator, maxillofacial surgeon, AZ Sint-Jan AV
Other Study IDs: 2368
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cleft Palate Children
Keywords: 3D virtual software; bone graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cleft patient requiring bone graft: Patients presenting at the division of maxillofacial surgery at the AZ Sint-Jan Brugge-Oostende av (Belgium) or the 1st department of pediatrics at the USemmelweis (Hungary) for bone graft surgery of the unilateral cleft receive a complete routine work-up, including a cone-beam CT (CBCT).

SUMMARY:
Objective: The investigators aim to compare the licensed Brainlab Iplan® software, considered the gold standard, to the 3D slicers and Blender freeware for the segmentation of the unilateral cleft defect, as well as the creation of individual 3D template for development of the bone graft.

Study design Retrospective, pilot study Patients presenting at the division of maxillofacial surgery at the AZ Sint-Jan Brugge-Oostende av (Belgium) or the 1st department of pediatrics at the USemmelweis (Hungary) for bone graft surgery of the unilateral cleft receive a complete routine work-up, including a cone-beam CT (CBCT). A single surgeon will run all the virtual planning steps with both the licensed software and the freeware. Timing of the four major steps will be measured with a digital chronometer (http://www.online-stopwatch.com/download-stopwatch/).

Ten children, 5 Belgian patients and 5 Hungarian patients, that already had a work-up and surgery for a unilateral cleft requiring a bone graft, will be planned. This based on the preoperative CBCT that is already present, by using both the licensed software and free software. The investigator will register patients' age, gender and cleft size and register the required time to complete the different planning steps, as well as list the number of actions to complete the planning, and the occurrence of software bugs. In addition, the learning effect will be examined through comparison of the different cases planned by the same surgeon. All patients will be planned twice with an interval of two weeks in order to measure intra-observer reliability. Moreover, a second surgeon will also plan the 10 cases to measure inter-observer reliability.

Main study endpoints The investigators hypothesize that the licensed software is more user-friendly, ensuring a significant shorter overall treatment planning time to create a model for accurate bone transfer from the iliac crest to the jawbone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a unilateral cleft
* Patients of all genders
* Patients aged 7-12 years old
* Patients should have presented themselves at the division of maxillofacial surgery, at the participating hospital centers, for bone graft surgery
* Patients should have received standardized cone-beam computed tomography (CBCT) image acquisition as part of routine work-up, and all original DICOM files should be present
* Preoperative 3D virtual planning should be performed by the same investigator per center with both the licensed software and the freeware

Exclusion Criteria:

* All patients that do not fit the abovementioned description
* Patients with previous bone graft surgery
* Patients with posttraumatic deformity
* Patients with preprosthetic indication

Ages: 7 Years to 12 Years | Sex: All
Age Groups: Child
Gender Based: Yes
Study Population: Patients presenting at the division of maxillofacial surgery at the AZ Sint-Jan Brugge-Oostende av (Belgium) or the 1st department of pediatrics at the USemmelweis (Hungary) for bone graft surgery of the unilateral cleft receive a complete routine work-up, including a cone-beam CT (CBCT).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
duration of total virtual planning time | preoperative
  measurement of total virtual planning time, with a digital chronometer

SECONDARY OUTCOMES:
duration of segmentation of the cleft defect | preoperative
  measurement of segmentation of the cleft defect, with a digital chronometer
duration of creation of the individual 3D template | preoperative
  measurement of duration of creation of the individual 3D template, with a digital chronometer

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium